CLINICAL TRIAL: NCT06089356
Title: Zolmitriptane as Prophylactic Therapy Childhood Migraine
Brief Title: Zolmitriptane as Prophylaxis for Chilhood Migraine
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Sherief Abd-Elsalam, professor, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Migraine
Record Dates: First submitted 2023-10-13; First posted 2023-10-18 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Topiramate; Valproic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- zolmitriptane (Active Comparator): zolmitriptane tablet daily
  Interventions: Drug: zolmitriptanee
- topiramate (Active Comparator): topiramate tablet daily
  Interventions: Drug: topiramate
- valproate (Active Comparator): valproate once daily
  Interventions: Drug: Valproate

INTERVENTIONS:
Drug: zolmitriptanee — zolmitriptane tablet daily
  Other Names: zolmitriptane tablet
  Arms: zolmitriptane
Drug: topiramate — topiramate once daily
  Other Names: topiramate tablet
  Arms: topiramate
Drug: Valproate — valproate once daily
  Other Names: Valproate tablet
  Arms: valproate

SUMMARY:
zolmitriptane can be tried as prophylactic therapy of childhood migraine

DETAILED DESCRIPTION:
90 children with migraine included in the study first group 30 received zolmitriptane second group 30 received topiramate third group 30 received valproate

ELIGIBILITY:
Inclusion Criteria:

children with migraine -

Exclusion Criteria:

those who suffer from ischemic heart disease , or who have allergy to any of drugs used

-

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
number and severity of migraine attacks | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Abeer Salamah, ass prof, Principal Investigator — kafrelsheikh university- egypt
Locations (1):
- Kafrelsheikh University, Tanta, Kafrelsheikh, Egypt

IPD SHARING:
Plan to Share IPD: No